CLINICAL TRIAL: NCT05699863
Title: A Multidisciplinary Approach to Screening for Obesity Complications - The MULTISITE Study
Brief Title: The MULTISITE Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Aase Handberg, Professor, Aalborg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-013
Record Dates: First submitted 2022-04-19; First posted 2023-01-26 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: NAFLD; Obesity; Extracellular Vesicles; Weight Loss
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: The study has three three groups, including obese (BMI 30,0 - 39,9 kg/m2) individuals (obese group) and lean (BMI 18,5 - 24,9 kg/m2) age and sex-matched control individuals (control group).
  Based on initial enrolment into the obese group, individuals with NAFLD (>5% hepatic steatosis) and metabolic syndrome (according to International Diabetes Foundation (IDF) consensus) will undergo a 4-5 month lifestyle intervention (intervention group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metabolically unhealthy obese (Intervention group) (Experimental): Obese (BMI: 30.0 - 39.9) participants with non-alcoholic fatty liver disease and metabolic syndrome.
  Interventions: Behavioral: Lifestyle intervention
- Metabolically healthy obese (Comparison group 1) (No Intervention): Obese individuals considered metabolically healthy based on them not presenting non-alcoholic fatty liver disease or metabolic syndrome.
- Healthy normal weight (Comparison group 2) (No Intervention): Normal weight individuals without non-alcoholic fatty liver disease or metabolic syndrome.

INTERVENTIONS:
Behavioral: Lifestyle intervention — Lifestyle intervention in the form of individualised dietitian consultation with the overall goal of weight loss.
  Intervention includes one initial consultation with a dietician of 1 hour and 15 minutes where participants receive a personalised diet-plan customised to the participants everyday life. After the initial consultation, the participants attend 10 "follow-ups" of about 25 minutes that are spread out over 4-5 months.
  Arms: Metabolically unhealthy obese (Intervention group)

SUMMARY:
This study will investigate potential correlations and relationships between obesity and organ-specific complications, including non-alcoholic fatty liver disease (NAFLD), non-alcoholic fatty pancreas disease (NAFPD) and fatty kidney. Furthermore, it will investigate how and if a lifestyle-induced weight-loss intervention decreases liver fat and improve NAFLD.

Furthermore, the study will investigate if extracellular vesicles (EVs) can be used as a biomarker for early detection of any of the above-mentioned by comparing obese individuals with NAFLD and metabolic syndrome with both normal weight controls and obese individuals without NAFLD and metabolic syndrome. Lastly, it will investigate if weight changes and the resulting improvement of NAFLD are accompanied by changes in liver-specific extracellular vesicle (EV) phenotypes.

DETAILED DESCRIPTION:
The worldwide prevalence of obesity and obesity-associated complications is increasing. A common feature associated with obesity is an increased ectopic and visceral fat inside and around the liver, kidney and pancreas. Ectopic and visceral fat is associated with systemic and local pathologies, including liver disease, pancreas disease, and kidney disease.

Current tools for diagnosis of obesity-related morbidities are insufficient, where methods either have low diagnostic accuracy, are too expensive, or invasive. This limits their use for patient care. Thus, there is a need for suitable non-invasive biomarkers for obesity-related complications that allow for screening, risk-stratification, and treatment evaluation of the growing obese population. In this context, extracellular vesicles (EVs) are of particular interest. EVs are small membrane-encapsulated particles released from cells into the blood circulation, and each EV can be considered a micro-biopsy of one single cell. It is proposed that differences in EV number and phenotype can function as potential biomarkers for obesity-related complications.

Early intervention against obesity and related complications minimizes future diseases. As obesity and its complications are associated with a positive energy balance, the best intervention is increased energy expenditure and/or decreased energy intake , leading to weight loss. Intervention against obesity requires permanent lifestyle changes, which can be helped by e.g., individualised diet and exercise plans, surgery, and counselling.

The aims of this project are thus, 1) to investigate visceral and ectopic fat and its associated complications with focus on NAFLD, NAFPD and fatty kidney. 2) investigate whether EVs can function as potential non-invasive biomarkers for any of these conditions, and 3) investigate if a lifestyle intervention decreases liver visceral and ectopic fat, and whether this improvement is reflected by an improvement of NAFLD and changes in EV phenotypes. The specific aims are as follows:

1. Investigate potential correlations and relationships between obesity and organ-specific complications, including NAFLD, NAFPD and fatty kidney;
2. Compare obese participants with lean control subjects, and investigate whether organ-specific EVs can be used as a biomarker for early detection of any of the above-mentioned conditions/states;
3. Investigate how and if a lifestyle-induced weight-loss intervention decreases liver fat and improve NAFLD. Furthermore, investigate if weight changes and the resulting improvement of NAFLD are accompanied by changes in liver-specific EV phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60
* BMI between 30,0 - 39,9 kg/m2.
* Signed informed consent.
* Metabolic syndrome
* NAFLD
* Wishes to participate in a weight reduction program.

Exclusion Criteria:

* Diabetes or any significant endocrine, heart, kidney, liver, or malignant disease.
* Pregnancy, planned pregnancy, or breast-feeding during the trial.
* Alcohol abuse or abuse of recreational drugs
* Medical treatment (systemic glucocorticoids, steatosis-inducing drugs, antibiotics up to two months prior to inclusion, or chemotherapy) or participation in clinical trials other than this.
* Excessive weight loss within the last three months (defined as more than 10 kilograms).
* Contraindications for MRI and dual energy x-ray absorptiometry (DEXA)scanning.
* Any medical condition or history thereof or any deviation from normal laboratory values that, in the opinion of the investigator, clinically contraindicates or hinders the completion of the trial procedures.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2036-01-31 (Estimated)

PRIMARY OUTCOMES:
Effect of weight loss on organ steatosis | 36 months
  Changes in steatosis of the liver, pancreas and kidneys assessed by magnetic resonance imaging (proton density fat fraction) between baseline, during weight loss, and after weight loss.
Effect of weight loss on plasma alanine transaminase | 36 months
  Changes in plasma alanine transaminase (IU/L) between baseline, during weight loss, and after weight loss.
Effect of weight loss on BMI | 36 months
  Changes in BMI between baseline, during weight loss, and after weight loss.
  Weight and height will be combined to report BMI in kg/m^2.
Effect of weight loss on total body fat | 36 months
  Changes in total body fat (%) as assessed by dual dual energy x-ray absorptiometry between baseline, during weight loss, and after weight loss.
Effect of weight loss on the homeostasis model assessment for insulin resistance | 36 months
  Changes in Homeostasis model assessment for insulin resistance (HOMA) between baseline, during weight loss, and after weight loss.
  Insulin (pmol/L) and plasma glucose (mmol/L) will be combined to calculate HOMA using the iterative structural model.
Effect of weight loss on plasma aspartate transaminase | 36 months
  Changes in plasma aspartate transaminase (IU/L) between baseline, during weight loss, and after weight loss.

SECONDARY OUTCOMES:
Extracellular vesicles as biomarkers in disease monitoring | 36 months
  Changes in extracellular vesicle concentration and phenotype assessed by high-resolution flow cytometry. Changes are defined as differences of extracellular vesicle concentrations and phenotypes between baseline, during weight loss, and after weight loss.
Extracellular vesicles as biomarkers for NAFLD diagnosis | 36 months
  Differences in extracellular vesicle concentration and phenotype assessed by high-resolution flow cytometry between participants with and without NAFLD.

CONTACTS AND LOCATIONS:
Overall Officials: Aase Handberg, Prof MD DMSc, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, North Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No
There is a general wish too share Individual Participant Data (IPD), however, due to stringent data and personal data protection considerations, it will not be possible unless data can be fully anonymised in the future.